CLINICAL TRIAL: NCT00226824
Title: Pilot Examination of Galantamine in the Management of Tic Disorders
Brief Title: Safety Study of Galantamine in Tic Disorders
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit subjects into the trial.
Sponsor: Parkinson's Disease and Movement Disorders Center (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAL-EMR-4017
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Tourette's Syndrome; Motor Tic Disorder; Vocal Tic Disorder
Keywords: Tourette's disorder; tic
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Tics | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine

SUMMARY:
The purpose of this study is to determine the safety, tolerability and efficacy of galantamine in tic disorders. The impact of galantamine on commonly associated behaviors (i.e. attention, obsessions, etc.) will also be examined.

DETAILED DESCRIPTION:
Modulation of cholinergic activity is a growing focus in neurologic therapeutics especially for dementing disorders such as Alzheimer disease. Treatment with the recently developed cholinesterase inhibitor, galantamine, has demonstrated significant improvement with few issues related to tolerability. In addition to inhibiting the activity of acetylcholinesterase, galantamine also modulates the activity of nicotinic cholinergic receptors by an allosteric mechanism. As a result, galantamine therapy may be beneficial when the response to other agents has been limited.

Cholinesterase inhibitor therapy has been reported to improve motor tics in children with TS refractory to more traditional therapies. Symptoms of co-morbid behavioral disorders, primarily inattention, were also improved. Cholinergic modulation appears a promising avenue for managing tic disorders.

Men and women (18 - 50 years of age) fulfilling DSM IV criteria for the diagnosis of chronic motor tic disorder, chronic vocal tic disorder or Tourette Syndrome and experiencing suboptimal control of tics on current therapy will be enrolled into this open label evaluation of galantamine. A total of 6 visits will be required over 22 weeks. Participants will follow a standard 4 week titration schedule achieving 12 mg bid after 8 weeks. They will maintain at 12 mg bid, or the maximum tolerated dose, for a further 8 weeks and then be withdrawn from therapy. The difference in tic severity prior to and upon completion of therapy will be examined. The impact of treatment upon obsessions/compulsions, attention/concentration, depression, anxiety and quality of life will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* DSM IV criteria for the diagnosis of Tourette's syndrome, chronic motor or chronic vocal tic disorder
* Accepted method of birth control

Exclusion Criteria:

* Preganancy or nursing
* Unstable medical illness
* Unstable psychiatric illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2005-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Treatment related adverse experience
Severity Score of the Yale Global Tic Severity Scale

SECONDARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Survey
Connors Adult Attention Deficit Hyperactivity Rating Scale
Hamilton Rating Scale for Depression
Hamilton Rating Scale for Anxiety
Short Form 36

CONTACTS AND LOCATIONS:
Overall Officials: Donald S Higgins, M.D., Principal Investigator — Parkinson's Disease and Movement Disorder Center of Albany Medical Center
Locations (1):
- Parkinson's Disease and Movement Disorders Center of Albany Medical Center, Albany, New York, United States

REFERENCES:
- [Background] Hoopes SP. Donepezil for Tourette's disorder and ADHD. J Clin Psychopharmacol. 1999 Aug;19(4):381-2. doi: 10.1097/00004714-199908000-00019. No abstract available. PMID 10440471
- [Background] Wilens TE, Biederman J, Wong J, Spencer TJ, Prince JB. Adjunctive donepezil in attention deficit hyperactivity disorder youth: case series. J Child Adolesc Psychopharmacol. 2000 Fall;10(3):217-22. doi: 10.1089/10445460050167322. PMID 11052411
- [Background] Hayslett RL, Tizabi Y. Effects of donepezil on DOI-induced head twitch response in mice: implications for Tourette syndrome. Pharmacol Biochem Behav. 2003 Dec;76(3-4):409-15. doi: 10.1016/j.pbb.2003.08.015. PMID 14643839
- [Background] Burt T. Donepezil and related cholinesterase inhibitors as mood and behavioral controlling agents. Curr Psychiatry Rep. 2000 Dec;2(6):473-8. doi: 10.1007/s11920-000-0005-7. PMID 11122998